CLINICAL TRIAL: NCT06116643
Title: Development of a Soluble Protein Hydrolysate (SPHi) as a Medical Food for the Treatment of Ulcerative Colitis
Brief Title: Pilot Study of a New Medical Food in the Management of Ulcerative Colitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Karl Sylvester, Professor-University Med Line, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-72442
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard Active Therapy plus SPHi (Experimental): Participants will undergo the standard active therapy of ulcerative colitis plus the addition of the ProGo medical food.
  Interventions: Dietary Supplement: Soluble protein hydrolysate (SPHi)

INTERVENTIONS:
Dietary Supplement: Soluble protein hydrolysate (SPHi) — Participants that are already on stable maintenance therapy for ulcerative colitis will continue with their therapy regimen and the addition of 10g of SPHi in 100ml of water every day for 12 weeks.

SUMMARY:
The goal of this clinical trial is to determine at how well a new medical food works in managing inflammation associated with ulcerative colitis in children. The main question it aims to answer is:

1) How well does the new medical food lower an inflammatory biomarker known as fecal calprotectin (fCal) in ulcerative colitis as compared to the historical active therapy levels of fCal? Participants will take a specified dose of the medical food in water each day for 12 weeks. The level of fCal will be measured through a stool sample at baseline, one during the 12 weeks, at the end of 12 weeks, and once more at 16 weeks. The levels of fCal will be compared across the 16 weeks and compared with levels before the new medical food was taken.

DETAILED DESCRIPTION:
The objective of this clinical trial is to assess the physiological response to a biologic food substance in maintenance therapy for ulcerative colitis in children. This will be measured through the measurement of fecal calprotectin (fCal) levels across the study period as well as in comparison to historical active therapy levels. Secondary endpoints will include a variety of biologic markers (inflammatory, microbial, metabolic) as well as clinical scores including patient reported outcomes and serum-based biomarkers such as ferritin and hemoglobin. The aim is to evaluate the effectiveness of the medical food as a safe and well-tolerated non-pharmacologic approach for reducing dependence on drug therapies and their associated side effects in the treatment of ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients with a confirmed diagnosis of ulcerative colitis on stable maintenance therapy.

Exclusion Criteria:

Pediatric patients with a confirmed diagnosis of ulcerative colitis who utilize oral or topical corticosteroids in maintenance therapy.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Fecal Calprotectin Levels | Enrollment through the post end of treatment follow-up at 16 weeks.
  Level of fecal calprotectin in stool sample at each study visit and compared to historical active therapy fecal calprotectin levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided